CLINICAL TRIAL: NCT07166198
Title: Mitigating Neural Hypoexcitability and Weakness During Disuse in Women
Acronym: MiND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Joshua Carr, Assistant Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12503; 5P20GM113109-09 (NIH)
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Muscle Weakness
Keywords: Resistance Training; Neuroplasticity; Muscle Disuse; Wrist immobilization; Women's Health
MeSH Terms: conditions — Muscle Weakness | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Two-phase, parallel-group randomized controlled design targeting midlife women aged 40-65 years, stratified by menopausal status.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention Group (TRAIN) (Experimental): This group will receive the experimental intervention
  Interventions: Device: Wrist immobilization; Behavioral: Resistance training; Behavioral: Resistance training rehabilitation
- Control Group (CON) (Active Comparator): This group will not receive the experimental intervention
  Interventions: Device: Wrist immobilization; Behavioral: Resistance training rehabilitation

INTERVENTIONS:
Device: Wrist immobilization — The wrist immobilization will use a medical device (wrist cast) to immobilize the left, non-dominant wrist for 7 days.
Behavioral: Resistance training — The cross-education intervention will consist of resistance training on the dominant, right hand.
  Arms: Intervention Group (TRAIN)
Behavioral: Resistance training rehabilitation — The resistance training rehabilitation will occur for the non-dominant, left hand following the immobilization phase for all participants.

SUMMARY:
Clinical trial The goal of this clinical trial is to learn how muscle weakness and atrophy develop during short periods of arm immobilization and whether a type of exercise called cross-education can help reduce these effects in women at midlife.

The main questions it aims to answer are:

What changes happen in the nervous system that lead to weakness when a wrist is immobilized?

Can training the opposite arm help maintain muscle strength, muscle size, and nervous system function in the immobilized arm?

Researchers will compare women who have their wrist immobilized with or without opposite-arm resistance training.

Participants will:

Wear a wrist cast on one arm for 7 days

Complete strength training with the opposite arm or no training, depending on their group

Attend study visits for strength and nervous system testing

Have non-invasive tests (like magnetic brain stimulation, muscle recordings, and muscle imaging) to measure how the nervous system and muscle responds

DETAILED DESCRIPTION:
This clinical trial employs a two-phase, parallel-group randomized controlled design targeting midlife women (ages 40-65), stratified by menopausal status. Participants will be randomized to either a cross-education training group (TRAIN) or a standard care control group (CONTROL).

Phase 1 (Immobilization and Cross-Education Intervention):

To induce rapid declines in neuromuscular function, participants will undergo unilateral wrist immobilization of the non-dominant arm using a hard cast for 7 days. During this period, the TRAIN group will complete three supervised resistance training sessions with the non-immobilized arm, while the CONTROL group will remain inactive. The intervention protocol emphasizes eccentric-biased resistance exercise, as prior data indicate that eccentric contractions optimize neural adaptation and mechanical loading. The protocol was developed from prior laboratory work and proof-of-concept interventions, with the goal of maximizing the cross-education response.

Phase 2 (Rehabilitation and Recovery):

Following cast removal, both groups will complete a 2-week standardized rehabilitation program (3 sessions per week) designed to restore wrist strength and function in the previously immobilized arm. Rehabilitation training is supervised and includes progressive resistance exercise to target recovery of neuromuscular performance.

ELIGIBILITY:
Inclusion Criteria:

* Women between 40-65 years of age
* Baseline handgrip strength >20Kg
* Right-hand dominant

Exclusion Criteria:

* Personal or family history of blood clots
* Current use of anticoagulant medications
* Neuromuscular or metabolic diseases (e.g., multiple sclerosis, diabetes)
* Arthritis
* Osteoporosis or osteopenia
* History of myocardial infarction within the past year
* Chronic pain ≥3/10 for ≥3 months
* Uncontrolled hypertension (≥140/90 mmHg)
* Upper extremity surgery within the past year
* Use of assistive hand or arm device within the past year
* Fall involving the upper extremities within the past year
* Upper extremity injuries preventing safe participation
* Use of body composition-altering medications (e.g., testosterone, GLP-1 agonists) in past 6 months
* Current use of muscle relaxants, benzodiazepines, or similar drugs
* Smoking within the past 6 months
* History of drug or alcohol abuse within the past year
* Severe anxiety or claustrophobia
* Pregnancy (current or planned)
* Allergies to medical adhesives
* High risk of sarcopenia (per SARC-F)
* Contraindications to TMS or MRI
* Not right-hand dominant
* Upper-body resistance training within the past 6 months
* Inability/unwillingness to refrain from resistance training during study

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Handgrip Strength | Baseline, immediately post-immobilization at 1 week, and post-rehabilitation at 3 weeks.
  Maximal handgrip strength (Kg) using an isometric handgrip dynamometer.
Wrist Extension Strength | Baseline, immediately post-immobilization at 1 week, and post-rehabilitation at 3 weeks.
  Peak torque (Nm) of the wrist extensor muscles measured using isokinetic dynamometry
Wrist Flexion Strength | Baseline, immediately post-immobilization at 1 week, and post-rehabilitation at 3 weeks.
  Peak torque (Nm) of the wrist flexor muscles measured using isokinetic dynamometry.

SECONDARY OUTCOMES:
Wrist Muscle Cross-Sectional Area and Volume (CT Imaging) | Baseline, immediately post-immobilization at 1 week, and post-rehabilitation at 3 weeks.
  Muscle cross-sectional area (cm²) and volume (cm³) of the wrist extensors and flexors, assessed using computed tomography (CT). Scans will be obtained at standardized anatomical landmarks of the forearm. Cross-sectional images will be segmented and analyzed with imaging software to quantify muscle size. The primary outcome is mean muscle cross-sectional area, with muscle volume derived from consecutive slices. These measures provide indices of muscle size and atrophy/hypertrophy over time.
Motor Evoked Potential (MEP) Amplitude | Baseline, immediately post-immobilization at 1 week, and post-rehabilitation at 3 weeks.
  Amplitude (mV) of motor-evoked potentials elicited by single-pulse TMS applied over the primary motor cortex of the left wrist and recorded from the extensor carpi radialis muscle. Larger amplitudes reflect greater corticospinal excitability.
Short-Interval Intracortical Inhibition (SICI) | Baseline, immediately post-immobilization at 1 week, and post-rehabilitation at 3 weeks.
  Short-interval intracortical inhibition assessed by paired-pulse TMS with a subthreshold conditioning stimulus followed by a suprathreshold test stimulus at an interstimulus interval of 2-5 ms. Outcome is the percent suppression of MEP amplitude relative to unconditioned trials.
Long-Interval Intracortical Inhibition (LICI) | Baseline, immediately post-immobilization at 1 week, and post-rehabilitation at 3 weeks.
  Assessed using paired-pulse TMS with a suprathreshold conditioning stimulus followed by a suprathreshold test stimulus at an interstimulus interval of 50-200 ms. LICI is quantified as the percent suppression of conditioned motor-evoked potential (MEP) amplitude relative to unconditioned MEPs.
Intracortical Facilitation (ICF) | Baseline, immediately post-immobilization at 1 week, and post-rehabilitation at 3 weeks.
  Assessed using paired-pulse TMS with a subthreshold conditioning stimulus followed by a suprathreshold test stimulus at an interstimulus interval of 8-20 ms. ICF is quantified as the percent increase of conditioned MEP amplitude relative to unconditioned MEPs.
Active Motor Threshold (AMT) | Baseline, immediately post-immobilization at 1 week, and post-rehabilitation at 3 weeks.
  Defined as the lowest TMS stimulus intensity (expressed as a percentage of maximum stimulator output) required to evoke MEPs ≥200 μV in at least 5 out of 10 consecutive trials during voluntary contraction of the target muscle at 10% of maximal effort. AMT reflects corticospinal excitability during an active state.

OTHER OUTCOMES:
Menopausal Hormone Profile | Baseline
  Serum concentrations of estradiol, luteinizing hormone (LH), and follicle-stimulating hormone (FSH) will be assessed from venous blood draws.
Physical Activity Levels | Phase 1 (1 week immobilization) and Phase 2 (2-3 weeks rehabilitation)
  Physical activity levels, including daily step count and energy expenditure will be assessed using triaxial accelerometers (ActiGraph wGT3X-BT) worn on the dominant wrist.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Carr, Ph.D., Principal Investigator — Kansas State University
Locations (1):
- Neuromuscular Physiology Laboratory, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results of publications (e.g., outcome measures, demographics, adverse events) will be deposited in a publicly accessible data repository (Open Science Framework). Data will be available following publication of primary results. Supporting materials, including the study protocol and statistical analysis plan, will also be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following publication of primary results.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan) will be available on the Open Science Framework (OSF) repository following publication of primary results. Data will be accessible to all registered OSF users without restriction. Users will be able to download the datasets and associated documentation directly from the project repository page.
URL: https://osf.io/registries?view_only=